CLINICAL TRIAL: NCT01598402
Title: Efficacy and Cost Efficacy of Prophylactic Treatment With Antibiotics During Concomitant Chemoradiotherapy in Patients With Locally Advanced Head and Neck Cancer to Prevent Aspiration Pneumonia. A Randomized Phase II-III Study
Brief Title: Efficacy of Prophylactic Treatment With Antibiotics During Concomitant Chemoradiotherapy in Patients With Head and Neck Cancer to Prevent Aspiration Pneumonia
Acronym: PANTAP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCNONCO201007
Record Dates: First submitted 2012-02-02; First posted 2012-05-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Head and Neck Cancer
Keywords: LAHNC; Locally Advanced Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No prophylactic treatment (No Intervention): When a lower airway infection is suspected cultures will be taken and a chest radiography will be made; after that the standard care will be given (in most patients admission to hospital and start of intravenous antibiotics).
- prophylactic treatment (Experimental): Administration of prophylactic amoxicillin/clavulanic acid suspension, 625 mg tid, start day 29 after the start of CRT until 14 days after the end of CRT. If a lower airway infection is suspected cultures will be taken and a chest radiography will be made; after that the standard care will be given (in most patients admission to hospital and start of intravenous antibiotics)
  Interventions: Drug: amoxicillin/clavulanic acid suspension

INTERVENTIONS:
Drug: amoxicillin/clavulanic acid suspension — 625 mg tid, start day 29 after the start of CRT until 14 days after the end of CRT
  Other Names: The total duration of the use of amoxicillin /clavulanic acid suspension will be between 20 and 27 days.
  Arms: prophylactic treatment

SUMMARY:
Patients with locally advanced head and neck cancer treated with chemo-radiotherapy have (during and shortly after this treatment) a high risk of developing pneumonia by aspiration. This pneumonia is often associated with a hospital admission and affects the quality of life.

The purpose of the study, is to determine whether prophylactic antibiotics may decrease the development of pneumonia. Prophylactic antibiotics means that there are no signs of pneumonia are already

DETAILED DESCRIPTION:
Concomitant chemoradiotherapy (CRT) is used in locally advanced head and neck cancer (LAHNC). It will be administered to patients for unresectable disease or for organ preservation as primary treatment. Furthermore, it can be used as postoperative treatment in case high risk recurrent disease is present. This treatment induces a high rate of acute toxicity, such as mucositis, dermatitis, dysphagia, anorexia, and pain. Swallowing dysfunction and aspiration are seen in a high proportion (30%-100%) of patients and with an immense impact on Quality of life (QoL).

Around half of the patients will develop an aspiration pneumonia during or shortly after the treatment.

Patients, who develop fever during concomitant chemoradiotherapy, are most of the time admitted in the hospital. In the differential diagnosis pneumonia is on the first place in all those patients. The standard diagnostic procedures consist of a chest X-ray and culture of the sputum and blood. Pneumonia can lead to mortality in this frail patient group.

The treatment of patients treated with chemoradiotherapy who develop fever and have a definite or suspected pneumonia, is administration of antibiotics, most frequently intravenous amoxicillin/clavulanic acid.

LAHNC patients who are smoking and/or with malnutrition are at the highest risk of getting a pneumonia during or after radiotherapy. Because smoking is one of the risk factors of developing head and neck cancer chronic obstructive pulmonary disease (COPD) is frequently present in this group. Also, COPD is a known risk factor for developing pneumonias.

Aspiration is seen in all primary sites of head and neck cancer, sometimes it is seen more frequently in patients with cancer of the larynx and hypopharynx. No data of prophylactic administration of antibiotics are available in LAHNC patients. However, a Cochrane review was published to assess the effects of prophylactic antibiotic regimens for the prevention of respiratory tract infections(RTIs) and overall mortality in adults receiving intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LAHNC which will be treated with CRT as discussed by a multidisciplinary team (i.e. a head and neck surgeon, a medical oncologist, and a radiation oncologist). This can be CRT as primary treatment or postoperative CRT.
* Written informed consent
* Expected adequacy of follow-up

Exclusion Criteria:

* Patients with pneumonia within the last 14 days before start of CRT
* Patients with other infections within the last 14 days within the last 14 days before start of CRT
* Patients with use of maintenance antibiotics
* Patients with antibiotic treatment within the last 14 days before start of CRT
* Patients with an allergy on amoxicillin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
the number of definite pneumonia and/ or suspected pneumonia | from day 1 of 1 CRT until 3,5 mnd after the last CRT
  Definite pneumonia:
  Evidence of pneumonia on chest radiography or 3 or more of the following:
  Sustained fever (temperature> 100 f [38°C]), Rales or rhonchi on chest auscultation Sputum Gram stain showing substantial leukocytes Sputum culture showing a respiratory pathogen
  Suspected pneumonia:
  At least 2 of the 4 following features are present, without evidence of pneumonia on chest radiography:
  Sustained fever (temperature> 100 f [38°C]) Rales or rhonchi on chest auscultation Sputum Gram stain showing substantial leukocytes Sputum culture showing a respiratory pathogen

SECONDARY OUTCOMES:
effects on Quality of Life | Baseline, Day 28 last day of CRT, 3,5 months after CRT
  to investigate the effects on QoL after prophylactic treatment with antibiotics
  Patients fill in the following questionnaires:
  QLQ-C30, EORTC H&N35, PSHHN, EQ-5D and the VAS, SF-36
Number and kind of positive blood cultures | from day 1 of 1 CRT until 3,5 mnd after the last CRT
number of admissions to hospital | from day 1 of 1 CRT until 3,5 mnd after the last CRT
Number of days of admission | from day 1 of 1 CRT until 3,5 mnd after the last CRT
Effects on mortality | from day 1 of 1 CRT until 3,5 mnd after the last CRT
  Mortality due to definite and/or suspected pneumonia
effects on mucositis: grade and duration | from day 1 of 1 CRT until 3,5 mnd after the last CRT
  Mucositis grade according to CTCAE v.4.0 and duration
side effects of amoxicillin/clavulanic acid | from day 1 of 1 CRT until 3,5 mnd after the last CRT
  side effects of amoxicillin/clavulanic acid
Effects on numbers and causative agents of infections at other sites | during follow up
  numbers and causative agents of infections at other sites during follow up (3.5 months after the end of CRT)

CONTACTS AND LOCATIONS:
Overall Officials: C. van Herpen, MD, Principal Investigator — University Medical Centre Nijmegen
Locations (6):
- Netherlands (6):
  - Ziekenhuis Rijnstate, Arnhem, Gelderland
  - University Medical Center Nijmegen st Radboud, Nijmegen, Gelderland
  - Medisch Centrum Alkmaar, Alkmaar
  - University Medical Centre Groningen, Groningen
  - Medisch centrum Leeuwarden, Leeuwarden
  - Academical Hospital Maastricht (AZM), Maastricht